CLINICAL TRIAL: NCT01698840
Title: An Evaluation of the Effects of Two Levels of Vitamin D in Infants Fed Preterm or Transitional Formula on Serum 25-Hydroxyvitamin D and Bone Status in Preterm Infants: A Double-Blind, Randomized Controlled Trial
Brief Title: Effect of Vitamin D in Diets of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Mead Johnson Nutrition (Industry); The Children's Nutrition Research Center (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-31433
Record Dates: First submitted 2012-09-24; First posted 2012-10-03 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Premature Infants
Keywords: Vitamin D; Transitional Formula
MeSH Terms: conditions — Premature Birth | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Nutrition (Experimental): Starting between post menstrual age (PMA) 34 0/7 to 38 6/7 weeks, infants in the Investigational Nutrition group will receive vitamin D drops that are added to transitional formula daily through hospital discharge and at home until the outpatient follow-up visit at 52 weeks PMA.
  Interventions: Dietary Supplement: Vitamin D
- Routine Nutrition (Placebo Comparator): Starting between post menstrual age (PMA) 34 0/7 to 38 6/7 weeks, infants in the Routine Nutrition group will receive placebo drops that are added to transitional formula daily through hospital discharge and at home until the outpatient follow-up visit at 52 weeks PMA.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Arms: Investigational Nutrition
Dietary Supplement: Placebo
  Arms: Routine Nutrition

SUMMARY:
Transitional formulas (22 kcal/oz) are recommended for infants less than 35 weeks gestation at birth. However, few data are available related to follow-up of infants receiving these formulas who were 28-34 weeks gestation at birth.

Primary hypothesis: Provision of supplemental vitamin D to a transitional formula will lead to higher serum 25-hydroxyvitamin D (25-OHD) levels and no infant with a serum 25-OHD less than 20 ng/mL when assessed at approximately 52 weeks post-menstrual age (PMA).

ELIGIBILITY:
Inclusion Criteria:

* Born at 28 0/7 to 34 6/7 weeks PMA and 1000-2250 g birth weight.
* Currently 34 0/7 to 38 6/7 weeks post-menstrual age at time of consent.
* Born at Texas Children's (including Pavilion for Women) or Methodist campus hospitals or transferred within 48 hours of birth.
* Care expected to be provided at one of these institutions until discharge home.
* Any initial feeding will be permitted, but expected to transition to primarily (80% of feeds or up to 2 breast milk feeds per day) infant formula by 38 6/7 weeks PMA or hospital discharge, whichever comes first.
* Able to tolerate 22 kcal/oz transitional formula and receive a volume of at least 130 mL/kg/day total feeding volume.
* No longer receiving any form of mechanical ventilation or diuretics. Low flow nasal cannula (< ¼ LPM) will be permitted if it is anticipated this will be discontinued before hospital discharge.

Exclusion Criteria:

* Bronchopulmonary dysplasia (BPD) requiring daily use of diuretics beyond 38 6/7 weeks PMA (or hospital discharge, whichever comes first) and > 22 kcal/oz concentration formula beyond 38 6/7 weeks PMA.
* Major congenital anomalies, history of proven Stage 2 or above NEC, or severe feeding intolerance.
* Caloric density greater than 22 kcal/oz.
* Higher order multiples (However, twins are acceptable. Twins will be randomized together. Only data from 1 twin picked at random will be used in the final analyses.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Serum 25-hydroxyvitamin D (25-OHD) level at 52 weeks post-menstrual age | Last 7 days of hospitalization and at 52 weeks post-menstrual age (PMA)

SECONDARY OUTCOMES:
Change from Baseline in Alkaline phosphatase activity at 52 weeks post-menstrual age | Last 7 days of hospitalization and at 52 weeks PMA

CONTACTS AND LOCATIONS:
Overall Officials: Amy h, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States